CLINICAL TRIAL: NCT02855372
Title: Impact of the Age Difference Between the Donor and Recipient on the Morbidity and Mortality After Lung Transplantation. Study on a National Multicenter Cohort (COLT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-39
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung transplanted patients
  Interventions: Procedure: Lung transplantation

INTERVENTIONS:
Procedure: Lung transplantation

SUMMARY:
It is commonly accepted that the characteristics of the organ donor impact on the future post transplant. In lung transplantation (LP), the defining characteristics of the "ideal" donor includes an age less than 55 years. However, before the pulmonary graft shortage with a corresponding mortality still too high waiting list, the lung graft acceptance criteria were reassessed permitting criteria "extension" ( "marginal" graft). And were grafted, depending on the urgency and accessibility problems in the registry of potential candidate, organs from donors aged 55 and older with quite comparable to those obtained from younger donors . Nevertheless, it is common practice that the grafts from older donors are more readily allocated to older candidates and the most severe, as many confounding factors to assess the real impact of donor age on post-transplant evolution on small cohorts.

The main goal of this study is to compare the survival of lung transplant patients depending on the age difference between donor and recipient.

The study will be conducted from a broad national cohort of lung transplant patients registered in COLT ( Lung Transplantation COhort). Established in September 2009, promoted by the University Hospital of Nantes, COLT involves 11 lung transplant centers authorized on French territory. It provides a standardized common longitudinal monitoring of the recipient from his transplant. Currently more than 1,000 patients included in this study are transplanted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients, included in COLT cohort, thus having given a signed written consent
* Who received a lung transplant

Exclusion Criteria:

* Lung transplanted patients in a context of national priority
* Lung transplanted patients who died within 3 months after the surgery
* Patients for whom it is a second lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent a lung transplantation
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Age difference in years between donor and recipient | 1 day
  The age difference will then be able to define two groups of patients:
  * 1 group with an age difference < 10 years
  * 1 group with an age difference > 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Hôpital Nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No